CLINICAL TRIAL: NCT03510923
Title: Selective Rather Than Routine Histopathological Examination Following Appendectomy and Cholecystectomy; the FANCY Study.
Brief Title: Selective Rather Than Routine Histopathological Examination Following Appendectomy and Cholecystectomy
Acronym: FANCY
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Willem A. Bemelman, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W17_328
Record Dates: First submitted 2018-04-18; First posted 2018-04-27 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Appendix; Appendectomy; Appendiceal Neoplasms; Gallbladder; Cholecystectomy; Gallbladder Neoplasms
Keywords: Appendix; Appendectomy; Gallbladder; Cholecystectomy; Neoplasms; Pathology; Selective; Routine
MeSH Terms: conditions — Appendiceal Neoplasms; Gallbladder Neoplasms; Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who underwent an appendectomy: Patients of all ages who underwent an appendectomy in the elective or non-elective setting.
  Interventions: Other: Inspection and palpation of the appendix
- Patients who underwent a cholecystectomy: Patients of all ages who underwent a cholecystectomy in the elective or non-elective setting.
  Interventions: Other: Inspection and palpation of the gallbladder

INTERVENTIONS:
Other: Inspection and palpation of the appendix — The removed appendix will be evaluated for tumours by the operating surgeon by visual inspection and digital palpation of the specimen. The appendix will not be opened. The surgeon will report his or her findings on a predefined scoring form: he or she will report all abnormalities and writes down whether he or she considers there is an indication for histopathological examination. Subsequently, all specimens will be sent for histopathological examination. Histopathological examination will be conducted according to the local protocol. In case of a neoplasm of the appendix, the treatment strategy is discussed and decided by the local multidisciplinary team. If an additional more extensive resection is decided to be appropriate, the specimens of the re-resection will be evaluated for the presence of remaining tumour tissue.
  Groups: Patients who underwent an appendectomy
Other: Inspection and palpation of the gallbladder — The removed gallbladder will be evaluated for tumours by the operating surgeon by visual inspection and digital palpation of the specimen. The gallbladder is opened in its length, without cutting the cystic duct, and is inspected and palpated. The surgeon will report his or her findings on a predefined scoring form: he or she will report all abnormalities and writes down whether he or she considers there is an indication for histopathological examination. Subsequently, all specimens will be sent for histopathological examination. Histopathological examination will be conducted according to the local protocol. In case of a neoplasm of the gallbladder, the treatment strategy is discussed and decided by the local multidisciplinary team. If an additional more extensive resection is decided to be appropriate, the specimens of the re-resection will be evaluated for the presence of remaining tumour tissue.
  Groups: Patients who underwent a cholecystectomy

SUMMARY:
The FANCY study will investigate whether a selective policy of histopathological examination of appendices and gallbladders based on the intraoperative findings of the surgeon is safe and cost-effective.

DETAILED DESCRIPTION:
Traditionally, all surgically removed appendices and gallbladders are sent to the department of pathology for histopathological examination. This is most likely not necessary in appendices and gallbladders that are not suspicious for a tumour when inspected visually or by palpation. If not detected by visual inspection or palpation, the tumour is usually of early stage and already treated with the resection of the organ. A policy of selective histopathological examination based on the intraoperative findings of the surgeon can probably reduce the amount of appendices and gallbladders that have to be examined by the pathologist, without a risk of undertreatment, with less risk of overtreatment and huge savings annually. In the FANCY study, a nationwide prospective multicenter observational cohort study, all appendices and gallbladders will be evaluated for tumours by visual inspection and palpation by the operating surgeon. The operating surgeon will report his or her findings and also write down whether he or she thinks there is an indication for histopathological examination. Subsequently, all specimens are sent to the pathologist for histopathological examination. Therefore, no aberrant findings will be missed due to this study. The prospective cohort can be compared through modelling to a hypothetical situation where appendices and gallbladders are only examined by the pathologist on indication. The primary outcome is the number of patients per 1000 examined appendices/gallbladders with a neoplasm requiring additional therapy benefitting the patient that would have been unnoticed in the policy of selective histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo an appendectomy or cholecystectomy in the elective or non-elective setting.

Exclusion Criteria:

* Primary indication for surgery: strong suspicion or proven malignancy in the appendix or gallbladder.
* Appendix or gallbladder removed as part of more extensive surgery, so-called incidental appendectomies or cholecystectomies.
* Patients included in the ACCURE trial (effect of appendectomy on ulcerative colitis).
* The presence of a gallbladder polyp of >10 mm on preoperative imaging.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are scheduled to undergo an appendectomy or cholecystectomy in one of the participating centers in The Netherlands.
Sampling Method: Probability Sample
Enrollment: 17380 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Unnoticed neoplasms requiring additional therapy benefitting the patient | 3 months
  Number of patients per 1000 examined appendices/gallbladders with a neoplasm requiring additional therapy benefitting the patient that would have been unnoticed in the policy of selective histopathological examination.
Costs | 3 months
  Costs of the policy with selective and with routine histopathological examination of the appendix/gallbladder.

SECONDARY OUTCOMES:
Malignancies | 2 weeks
  Incidence of malignancies in resected appendices and gallbladders
Unnoticed malignancies | 2 weeks
  Incidence of unnoticed malignancies in resected appendices and gallbladders
Malignancies requiring more extensive resection or other additional treatment | 3 months
  Incidence of malignancies in resected appendices and gallbladders that subsequently require more extensive resection or other additional treatment.
Benefit of additional resection | 2 weeks
  Remaining tumour tissue and/or positive lymph nodes in re-resection specimen
Harm of additional resection | 1 month
  Incidence of postoperative complications
Other aberrant findings | 2 weeks
  Incidence of other aberrant findings as parasite infections, endometriosis, granulomatosis and benign neoplasms.
Other aberrant findings requiring additional therapy | 3 months
  Incidence of other aberrant findings as parasite infections, endometriosis, granulomatosis and benign neoplasms that require additional therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Willem Bemelman, Professor, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam-Zuidoost, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bastiaenen VP, Corten BJ, de Savornin Lohman EA, de Jonge J, Kraima AC, Swank HA, van Vliet JL, van Acker GJ, van Geloven AA, In 't Hof KH, Koens L, de Reuver PR, van Rossem CC, Slooter GD, Tanis PJ, Terpstra V, Dijkgraaf MG, Bemelman WA. Safety and cost analysis of selective histopathological examination following appendicectomy and cholecystectomy (FANCY study): protocol and statistical analysis plan of a prospective observational multicentre study. BMJ Open. 2019 Dec 23;9(12):e035912. doi: 10.1136/bmjopen-2019-035912. PMID 31874901